CLINICAL TRIAL: NCT03282747
Title: Risk Factors for Venous Thrombosis and Pulmonary Embolism in Blood Donors
Brief Title: Distribution of Risk Factors for Venous Thromboembolism in Blood Donors
Acronym: ANEMONE
Status: Completed | Type: Observational
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: University of Bari (Other)
Responsible Party: Principal Investigator, Elvira Grandone, MD, Head of Unit, MD, Casa Sollievo della Sofferenza IRCCS
Other Study IDs: ANEMONE/01
Record Dates: First submitted 2017-09-10; First posted 2017-09-14 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Venous Thromboembolism; Risk Factor, Cardiovascular; Blood Type
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: no intervention — no intervention

SUMMARY:
Venous thromboembolism occurs with an incidence of about 1 per 1000 per year in adults . The main consequences are death, recurrence, post-thrombotic syndrome and major bleeding due to anticoagulation. Mortality rates are lower among patients with idiopathic venous thrombosis and higher among those in whom thrombosis occurs in the presence of cancer.

The risk increases with the age for unclear reasons. There are also differences in the incidence according to ethnicity; however, data in subjects of European ancestry are scarce.

Several studies have documented an association between thrombosis and ABO group. Specifically, non-O blood groups have a higher risk of myocardial infarction, angina, peripheral vascular disease, cerebral ischemia and venous thromboembolism than O. While there are numerous studies carried out in patients who have already shown thromboembolic events, data on the incidence of risk factors in the healthy population are completely inadequate.

Understanding the risk factors for venous thrombosis is necessary to maximize the prevention of this disease in individuals and groups of high-risk patients . For this purpose a self-administered questionnaire will be used. Data obtained by blood donors on exposure to risk factors will be used to set up a clinical score to validate in future studies to carry out in patients with VTE.

DETAILED DESCRIPTION:
Venous thromboembolism, defined by deep vein thrombosis (DVT) and / or pulmonary embolism (PE), occurs with an incidence of about 1 per 1000 per year in adult populations. Rates are slightly higher in men than women. About two-thirds of the episodes are manifested as DVT and one third as PE with or without DVT. The main consequences of venous thrombosis are death, recurrence, post-thrombotic syndrome and major bleeding due to anticoagulation. Thrombosis is also associated with impaired quality of life, especially when developing posttrombotic syndrome. The mortality rate within one month from an episode is about 6% in patients with DVT and 10% in those with PE. The mortality rate for PE was estimated to be around 30% in the studies that included the PE diagnosis of autopsy, pointing out that many PEs are not clinically recognized before death. Mortality rates are lower among patients with idiopathic venous thrombosis and higher among those in whom thrombosis occurs in the presence of cancer.

Venous thrombosis is a most frequent disease in elderly patients with a low rate of about 1 per 10,000 per year before the fourth decade of life, which increases rapidly after the age of 45 and approaches 5-6 per 1000 per year at the age of 80 years. In a study, the rate of events over a period of 8 years and in individuals over 85 years of age was 13 times greater than that of individuals between 45 and 55 years, with an absolute rate of 7 per 1000 per year and a greater mortality in older people. It is likely that thrombosis is less diagnosed in some debilitated elderly patients so that these estimates are probably underestimated. The reasons for an increased risk of thrombosis with age are not clear, but may include the increasing presence of other thrombotic diseases, increased coagulation potential, or some combination of these.

There are also differences in the incidence of venous thrombosis diagnosed among lower-rate ethnic groups in the United States, Asians, Pacific Islanders, and Hispanics than Whites and with some studies showing an approximate rate of 25% higher in Afro-Americans. There is little information on the epidemiology of thrombosis in Europe.

Several studies have documented an association between thrombosis and ABO group. Specifically, non-O blood groups have a higher risk of myocardial infarction, angina, peripheral vascular disease, cerebral ischemia and venous thromboembolism (VTE) than O, probably because factor VIII, factor von Willebrand is lower in group 0 patients. While there are numerous studies conducted on patients who have already shown thromboembolic events, data on the incidence of risk factors in the healthy population are completely inadequate.

Understanding the risk factors for venous thrombosis is necessary to maximize the prevention of this disease in individuals and groups of high-risk patients . For this purpose blood donors will be requested to fill in a self-administered questionnaire. Healthy blood donors will be requested to give personal and family information regarding previous use of current of anticoagulant drugs, surgery, contraceptive use, pregnancy, previous blood transfusion. The presence of one or more risk factors will be used to set up a clinical score to validate in future studies on patients with previous VTE.

ELIGIBILITY:
Inclusion Criteria:

* Blood donors

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Blood donors consecutively observed
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Distribution of risk factors in blood donors | 1 year
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Casa Sollievo della Sofferenza, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No